CLINICAL TRIAL: NCT01765504
Title: Pilot Study of the Feasibility of Multicenter NIRS Data Collection and Interventions for Desaturation in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: Multicenter NIRS Study
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Disease
Keywords: Cardiac surgery; near infrared spectroscopy
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Using the 9 centers (Appendix B) involved with the planned multicenter NIRS comparative effectiveness trial the specific aims of this study are:

1. To demonstrate the feasibility of collecting rScO2 data from patients undergoing cardiac surgery in a multicenter study design.
2. To demonstrate the feasibility of using a standard algorithm for treating rScO2 desaturations during cardiac surgery in a multicenter study design.

DETAILED DESCRIPTION:
Brain injury after cardiac surgery is a chief source of patient mortality and healthcare costs and can significantly impair quality of life. Reducing the burden of this complication has wide public health implications. The broad manifestations of perioperative brain injury include stroke, delirium, and cognitive decline.5 All forms of injury are believed to result primarily from cerebral embolism and/or reduced cerebral blood flow (CBF). The risk for cerebral hypoperfusion is likely the highest during cardiopulmonary bypass (CPB), when mean arterial pressure (MAP) is kept low (~60 mmHg), particularly for patients who are aged and who have cerebral vascular disease. Near-infrared spectroscopy (NIRS) is used increasingly to monitor regional cerebral oxygen saturation (rScO2) in patients undergoing cardiac surgery, although limited data show that it improves patient outcomes. Regardless, clinical evidence supporting the efficacy of NIRS-based monitoring is needed urgently because the cost of NIRS sensors (~$220/patient) could add $132 million annually to hospital costs for cardiac surgery. We must address this issue quickly because the rising prevalence of NIRS use and advocacy by experts and industry will likely soon result in NIRS becoming a standard of care. We are in the process of submitting a multicenter, prospectively randomized comparative effectiveness trial to assess the efficacy of NIRS monitoring in patients who are undergoing coronary artery bypass graft (CABG) surgery with CPB, and/or valve surgery, and who are at risk for brain injury. The goal of the planned proposal is to determine whether interventions to correct rScO2 desaturations (value <50% or 20% reduction from room air baseline) reduce the frequency of neurologic and other complications compared with standard care (no clinical monitoring). In order to demonstrate feasibility of our proposal we need to demonstrate the ability of the team to collect rScO2 data from multiple centers and to show the ability of the team to properly follow an algorithm for treating rScO2 desaturations that occur during surgery. Thus, the aim of the current study is to collect preliminary data to support our larger comparative effectiveness trial.

ELIGIBILITY:
Inclusion Criteria: Patient inclusion criteria will be male or female patients >50 years of age undergoing primary or re-operative CABG and/or cardiac valve surgery that requires CPB who will have NIRS monitoring for clinical indications.

-

Exclusion Criteria: Emergency surgery

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient inclusion criteria will be male or female patients >50 years of age undergoing primary or re-operative CABG and/or cardiac valve surgery that requires CPB who will have NIRS monitoring for clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
rScO2 desaturation data collection | During Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Hogue, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Steppan J, Hogue CW Jr. Cerebral and tissue oximetry. Best Pract Res Clin Anaesthesiol. 2014 Dec;28(4):429-39. doi: 10.1016/j.bpa.2014.09.002. Epub 2014 Sep 28. PMID 25480772
- See also: http://www.meddium.com/charleshogue — http://www.meddium.com/charleshogue